CLINICAL TRIAL: NCT03430765
Title: Preventing Persistent Pain and Reducing Depressive and Anxious Symptoms Following Mastectomy and Lumpectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Hadlandsmyth (Other)
Collaborators: Holden Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Katherine Hadlandsmyth, Clinical Assistant Professor of Anesthesia - Chronic Pain Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201502709
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Persistent Postsurgical Pain; Breast Cancer Female; Ductal Carcinoma in Situ
MeSH Terms: conditions — Pain, Postoperative; Carcinoma, Intraductal, Noninfiltrating | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Standard breast cancer treatment plus a single 2 hour individual Acceptance and Commitment Therapy coping skills session.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as Usual (No Intervention): Standard breast cancer treatment.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Single 2-hour individual Acceptance and Commitment Therapy coping skills session.
  Arms: Acceptance and Commitment Therapy

SUMMARY:
The proposed study will be a pilot randomized controlled trial comparing treatment as usual (TAU) to treatment as usual plus a brief Acceptance and Commitment Therapy (ACT) intervention (TAU + ACT) with mastectomy and lumpectomy patients identified as at-risk for developing persistent post-operative pain. The ACT intervention is a single individual therapy session scheduled two weeks following surgery. Potential participants will be recruited from the University of Iowa Breast Cancer Clinic. A sample size of n = 30 for each arm will be recruited. An attrition rate of 20% is anticipated so the total N to be recruited for the study is 72 participants. Study measures will consist of self-report questionnaires and medical record data. Data will be collected prior to surgery, one-week after surgery, and 3 months after surgery.

DETAILED DESCRIPTION:
Psychological interventions addressing depression, anxiety, and psychological approaches to pain management in pre-surgical patients may serve to prevent the development of persistent post-surgical pain, depression, and anxiety in at-risk individuals. Acceptance and Commitment Therapy (ACT) is a psychological therapy that has been shown to be effective in minimizing the impairing impact of chronic pain and in treating depression and anxiety. ACT is a behavior therapy incorporating mindfulness, which aims to increase psychological flexibility via facilitating psychological acceptance and committed action in the direction of one's personally identified values. ACT has also shown promise in brief interventions, including a one day ACT workshop with patients with comorbid migraine and depression. The current study proposes to identify pre-operative breast cancer patients who are at increased risk for developing persistent post-surgical pain and to offer a brief ACT intervention with the aim of reducing the incidence of persistence post-surgical pain and psychological sequela.

ELIGIBILITY:
Inclusion criteria: 1) ≥18 years of age, 2) scheduled for mastectomy or lumpectomy for breast cancer or DCIS, 3) identified to be "at risk" (per guidelines below).

At risk criteria: Psychological distress (elevated anxiety, depression, or pain catastrophizing), under the age of 50, or with a pre-existing chronic pain condition. Scores of 10 or above on the Generalized Anxiety Disorders 7-item scale or the Personal Health Questionnaire Depression 8 item Scale will indicate elevated anxiety or depression. A score of 30 or above on the Pain Catastrophizing Scale will indicate elevated catastrophizing.

Exclusion Criteria:

1) language or cognitive barriers preventing completion of questionnaires, 2) severe psychiatric disorder: bipolar or psychotic disorder, 3) significant surgical complications.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06-21 (Actual); Primary Completion 2017-11-19 (Actual); Study Completion 2017-11-22 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | 3-months following surgery
  Surgical site pain severity (0 = no pain - 10 = pain as bad as you can imagine)

SECONDARY OUTCOMES:
The Brief Pain Inventory (BPI: pain severity) | 3-months following surgery
  Pain severity: four items: Average pain, worst in 24 hours, least in 24 hours, and right now (on a 0-10 scale)
The Brief Pain Inventory (BPI: pain interference) | 3-months following surgery
  Pain interference: 7 items rated on 0= does not interfere to 10 = completely interferes
Generalized Anxiety Disorder 7-item scale | 3-months following surgery
  Anxiety: score ranges from 0 (low anxiety) to 21 (high anxiety)
Patient Health Questionnaire -8 item | 3-months following surgery
  Depression: scores range from 0 (low depression) to 24 (high depression)
SF-12 Health Survey | 3-months following surgery
  Quality of Life: There are two subscales on this 12-item measure: the physical component summary and the mental component summary. Scores range from 0-100 with higher scores indicating better health.
Pain catastrophizing Scale | 3-months following surgery
  Pain catastrophizing: scores range from 0 (low catastrophizing) to 52 (high catastrophizing)
Chronic Pain Acceptance Questionnaire | 3-months following surgery
  Pain Acceptance: This 20 item scale has two subscales: Activity engagement (11 items) and Pain willingness (9 items), and a combined total score. Each item is rated on a scale of 0 -6. Higher scores indicate higher levels of acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hadlandsmyth, Ph.D., Principal Investigator — University of Iowa Hospital and Clinics
Locations (1):
- University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dindo L, Recober A, Marchman JN, Turvey C, O'Hara MW. One-day behavioral treatment for patients with comorbid depression and migraine: a pilot study. Behav Res Ther. 2012 Sep;50(9):537-43. doi: 10.1016/j.brat.2012.05.007. Epub 2012 May 27. PMID 22728646
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Powers MB, Zum Vorde Sive Vording MB, Emmelkamp PM. Acceptance and commitment therapy: a meta-analytic review. Psychother Psychosom. 2009;78(2):73-80. doi: 10.1159/000190790. Epub 2009 Jan 14. PMID 19142046
- [Background] Vowles, K.E., Wetherell, J.L., Sorrell, J.T. Targeting acceptance, mindfulness, and values-based action in chronic pain: Findings of two preliminary trials of an outpatient group-based intervention. Cognitive and Behavioral Practice 16: 49-58. 2009